CLINICAL TRIAL: NCT03913689
Title: A Prospective, Open-label, Long-term, Multi-center, Registry to Assess the Safety and Efficacy of the Bioness StimRouter Neuromodulation System in Subjects With Chronic Pain of Peripheral Nerve Origin
Brief Title: StimRouter Registry Clinical Protocol
Status: Completed | Type: Observational
Sponsor: Bioness Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-00001
Record Dates: First submitted 2019-03-25; First posted 2019-04-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Peripheral Neuropathy; Nervous System Diseases; Peripheral Nervous System Diseases; Peripheral Nervous System Problem; Peripheral Nerve Injuries; Peripheral Nervous
Keywords: peripheral nerve stimuation (PNS)
MeSH Terms: conditions — Chronic Pain; Peripheral Nervous System Diseases; Nervous System Diseases; Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- StimRouter Neuromodulation System: Implant of the Bioness StimRouter Neuromodulation System in subjects with chronic pain of peripheral nerve origin
  Interventions: Device: StimRouter Neuromodulation System

INTERVENTIONS:
Device: StimRouter Neuromodulation System — An implantable neuromodulation device that treats chronic peripheral nerve pain.

SUMMARY:
This Registry study will prospectively evaluate the long-term effectiveness, safety, and tolerability of the StimRouter Neuromodulation System, along with evaluating the technical performance of StimRouter, surgical outcomes, health-related quality of life, concomitant medical use, and subject's impression of improvement.

DETAILED DESCRIPTION:
This is a prospective, open-label, long-term, multi-center registry. Up to 173 subjects with chronic pain related to peripheral nerve will be enrolled by approximately 15 qualified sites. Subjects who are eligible for a StimRouter will be enrolled in order to evaluate the subject's experience at pre-implant, the implant, and post-implant for up to 24 months. Based on routine care, subjects will be seen at day of implant, within 2 weeks post-implant, 3 months post-implant, 6 months post-implant, 9 months post implant, 12 months post-implant, and 24 month post-implant.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age at the time of giving informed consent.
2. Subject who has chronic pain of peripheral nerve origin
3. Subject is eligible for StimRouter as determined by the Clinician.
4. Subject has a score of 5 or higher on the Pain NRS for average pain specific to the area(s) of chronic pain being treated over the past 24 hours
5. Subject is planned to be scheduled for implant of StimRouter.
6. Subject has a life expectancy greater than 6 months as determined by the Clinician.
7. Subject who is able to read, understand, and voluntarily sign the IRB-approved informed consent form prior to the performance of any study-specific procedures.
8. Subject who is able to understand and complete required assessments.

Exclusion Criteria:

1. Subject has other concomitant treatment or medical condition that, in the opinion of the Clinician, prevents the subject from study participation.
2. Subject who, for implantation in the trunk, has an implanted demand-type cardiac pacemaker or defibrillator.
3. Subject has or plans to have a Spinal Cord Stimulator (SCS), Peripheral Nerve field Stimulation System (PNfS), Dorsal Root Ganglion system (DRG), or implantable infusion pump.
4. Subject who has an implanted device in the area for StimRouter implantation without sponsor approval. Maintain a minimum separation distance of 6 inches (15 cm) between the StimRouter system and all other active implanted devices.
5. Subject who requires, or is likely to require, diathermy at the implant site.
6. Subject who requires, or is likely to require, therapeutic ultrasound at the implant site.
7. Subject who has a cancerous lesion present near the target stimulation point.
8. Subject with a bleeding disorder, which, in the opinion of the investigator, is a contraindication to device placement.
9. Subject who has an active systemic infection.
10. Subject who is immunocompromised and/ or determined by the Clinician to be clinically inappropriate for the procedure and implant.
11. Subject who has an active or existing skin disorder or irritation, which, at the Clinician's discretion, precludes the use of skin gel electrodes.
12. Subject who currently require or is likely to require Magnetic Resonance Imaging (MRI) within the MRI exclusion zone: the entire StimRouter lead must be at least 50 cm from the center of the MRI system's bore (the iso-center) and at least 16 cm outside of the MRI coil measured from the edge of the MRI coil.
13. Subject who has a history of adverse reactions to local anesthetic (e.g., lidocaine).
14. Subject who is pregnant, plan on becoming pregnant, or is breastfeeding during the study period.
15. Subject who is participating in any other study that could affect the outcome of the registry, such as a spinal stimulation study.
16. Subject who is in litigation related to their pain, or who has a pending or active worker's compensation claim. (A patient receiving long-term medical care from a settled Worker-s Compensation claim would not be excluded.)
17. Subject who declines to provide written consent or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 173 adult subjects (18 years or older) who have chronic pain of peripheral nerve origin, or other causes for which the Clinician determines StimRouter is the appropriate therapy.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain from Screening through 6 Months | Month 6
  Change from baseline to 6 months post-permanent implant in aversge pain assessed by using a Numeric Rating Scale

SECONDARY OUTCOMES:
Change in Pain Severity post-implantation | Month 6
  Average change from baseline to month 6 post-implantation in Pain Severity score as measured through the BPI-SF
Change in Pain Interference post-implantation | Month 6
  Average change from baseline to month 6 post-implantation in Pain Interference score as measured through the BPI-SF
Change in Health-related Quality of Life | MOnth 6
  Average change from baseline to month 6 in health-related quality of life as assess by the VR-12 questionnaire
Change in Patient Global Impression of change | Month 6
  Average change from baseline to month 6 in patient global impression of change (PGIC)
Patient Treatment Satisfaction | Month 6
  Overall patient treatment satisfaction survey
Pain medication use | Month 6
  Decrease in chronic pain related medication intake at month 6 when compared to baseline

OTHER OUTCOMES:
Change in average pain | Month 12
  Average change from baseline to Month 12 post-implantation measured through a NPRS scale
Change in average pain | Month 24
  Average change from baseline to Month 24 post-implantation measured through a NPRS scale
Change in Pain Severity | Month 12
  Average change from baseline to Month 12 post-implantation in Pain Severity measured through the BPI-SF
Change in Pain Severity | Month 24
  Average change from baseline to Month 24 post-implantation in Pain Severity measured through the BPI-SF
Change in Pain Interference | Month 12
  Average change from baseline to Month 12 post-implantation in Pain Interference measured through the BPI-SF
Change in Pain Interference | Month 24
  Average change from baseline to Month 24 post-implantation in Pain Interference measured through the BPI-SF
Change in Health-related Quality of Life | Month 12
  Average change from baseline to month 12 in health-related quality of life as assess by the VR-12 questionnaire
Change in Health-related Quality of Life | Month 24
  Average change from baseline to month 24 in health-related quality of life as assess by the VR-12 questionnaire
Change in Patient Global Impression of Change | Month 12
  Average change from baseline to month 12 in patient global impression of change (PGIC)
Change in Patient Global Impression of Change | Month 24
  Average change from baseline to month 24 in patient global impression of change (PGIC)
Pain Medication Use | Month 12
  Decrease in chronic pain related medication intake at month 12 when compared to baseline
Pain Medication Use | Month 24
  Decrease in chronic pain related medication intake at month 24 when compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Keith McBride, Study Chair — Bioness Inc; Eric Grigsby, MD, Study Director — Bioness Inc
Locations (9):
- United States (9):
  - University of California San Diego, La Jolla, California
  - California Orthopedics & Spine, Larkspur, California
  - Stanford University, Redwood City, California
  - Stamford Hospital, Stamford, Connecticut
  - International Spine,Pain and Performance Center, Washington D.C., District of Columbia
  - Warner Orthopedics, Baton Rouge, Louisiana
  - Albert Einstein/Moss Rehab, Elkins Park, Pennsylvania
  - Valley Sports and Spine Clinic, Blacksburg, Virginia
  - Advocate Aurora Health, Oshkosh, Wisconsin

IPD SHARING:
Plan to Share IPD: No